CLINICAL TRIAL: NCT02681211
Title: A Randomized Trial Comparing Auricular Acupuncture and Intravenous Migraine Medications in the Treatment of Status Migrainosus in the Pediatric Emergency Department
Brief Title: Auricular Acupuncture vs SOC in Migraine HA
Acronym: MigAcu
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Danielle Graff, Associate Professor, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15.0827
Record Dates: First submitted 2016-02-04; First posted 2016-02-12 (Estimated); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Migraine Headache
Keywords: migraine headache; acupuncture
MeSH Terms: conditions — Migraine Disorders | interventions — Acupuncture, Ear; Ketorolac; MAX protein, human; Ketorolac Tromethamine; Metoclopramide; Diphenhydramine; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Auricular Acupuncture (Experimental): If assigned to the auricular acupuncture arm, efficacious ear points will be located by a needle contact test and/or an electrical point finder which emits an acoustic alarm when a change in electrical resistance is detected signifying a potential active auricular acupoint.
  Interventions: Other: Auricular Acupuncture
- Medication and Fluid (Active Comparator): If assigned to receive intravenous medications and fluid the subject will be treated with the ED standard of care medications which include:
  1. Ketorolac 0.5mg/kg, max 30mg
  2. Metoclopramide 0.1 mg/kg, max 10mg
  3. Diphenhydramine 1mg/kg, max 50mg
  4. Normal saline fluid bolus 20mL/kg, max 1000mL
  Interventions: Drug: Ketorolac 0.5mg/kg, max 30mg; Drug: Metoclopramide 0.1 mg/kg, max 10mg; Drug: Diphenhydramine 1mg/kg, max 50mg; Drug: Normal saline fluid bolus 20mL/kg, max 1000mL

INTERVENTIONS:
Other: Auricular Acupuncture — ASP (acupuncture semi-permanent) gold needles will be placed in the efficacious ear points with a maximum of 3 needles in each ear.
  Arms: Auricular Acupuncture
Drug: Ketorolac 0.5mg/kg, max 30mg — If assigned to receive intravenous medications and fluid the subject will be treated with the ED standard of care medications which include:
  1. Ketorolac 0.5mg/kg, max 30mg
  2. Metoclopramide 0.1 mg/kg, max 10mg
  3. Diphenhydramine 1mg/kg, max 50mg
  4. Normal saline fluid bolus 20mL/kg, max 1000mL
  Other Names: Toradol
  Arms: Medication and Fluid
Drug: Metoclopramide 0.1 mg/kg, max 10mg — If assigned to receive intravenous medications and fluid the subject will be treated with the ED standard of care medications which include:
  1. Ketorolac 0.5mg/kg, max 30mg
  2. Metoclopramide 0.1 mg/kg, max 10mg
  3. Diphenhydramine 1mg/kg, max 50mg
  4. Normal saline fluid bolus 20mL/kg, max 1000mL
  Other Names: Reglan
  Arms: Medication and Fluid
Drug: Diphenhydramine 1mg/kg, max 50mg — If assigned to receive intravenous medications and fluid the subject will be treated with the ED standard of care medications which include:
  1. Ketorolac 0.5mg/kg, max 30mg
  2. Metoclopramide 0.1 mg/kg, max 10mg
  3. Diphenhydramine 1mg/kg, max 50mg
  4. Normal saline fluid bolus 20mL/kg, max 1000mL
  Other Names: Benadryl
  Arms: Medication and Fluid
Drug: Normal saline fluid bolus 20mL/kg, max 1000mL — If assigned to receive intravenous medications and fluid the subject will be treated with the ED standard of care medications which include:
  1. Ketorolac 0.5mg/kg, max 30mg
  2. Metoclopramide 0.1 mg/kg, max 10mg
  3. Diphenhydramine 1mg/kg, max 50mg
  4. Normal saline fluid bolus 20mL/kg, max 1000mL
  Other Names: Normal Saline
  Arms: Medication and Fluid

SUMMARY:
Patients with migraine headache will be offered the opportunity to participate in this randomized study evaluating auricular acupuncture versus standard treatment for migraine headaches for patients in the pediatric emergency department (ED).

DETAILED DESCRIPTION:
Potential subjects will be identified using the diagnosis of migraine headache classified by the modified ICHD-II (International Classification for Headache Disorders) criteria proposed by Hershey et. al. This diagnosis will be confirmed by the investigators prior to enrollment of the subject and will be documented in the study documents. Subjects will be recruited during the scheduled work or research hours of the investigators in the ED.

Eligible patients will be informed of the study including a discussion of the two possible interventions. After informed consent and assent are obtained, patients will be randomly assigned 1 of the 2 arms of the study. The target is 40 subjects in each arm. Subjects will be assigned to a study group using a computer generated randomization schema. This randomization will only be known to one unblinded collaborator that will not be enrolling subjects or be involved in the data analysis.

If assigned to receive intravenous migraine medications the subject will be treated with the standard of care medications which include ketorolac (0.5mg/kg, max 30mg), metoclopramide (0.1 mg/kg, max 10mg), diphenhydramine (1mg/kg, max 50mg) plus a normal saline fluid bolus (20mL/kg, max 1000mL).

If assigned to the auricular acupuncture arm, efficacious ear points will be located by a needle contact test and/or an electrical point finder which emits an acoustic alarm when a change in electrical resistance is detected signifying a potential active auricular acupoint. If the subject does not improve with acupuncture, they will be assessed by the ED physician and at the MD discretion further emergency department treatment will be administered which may include intravenous migraine medications as this is the current standard of care in the Norton Children's Hospital/Norton Children's Medical Center (KCH/KCMC) ED.

All subjects will be contacted 2 to 6 days after discharge to determine their clinical status. If the darts are still in place at the follow-up call, the subjects will be contacted at 2 weeks and weekly thereafter until all darts have fallen out.

ELIGIBILITY:
Inclusion Criteria:

* Confirmation of the diagnosis of migraine headache

Exclusion Criteria:

* Patients who received ED migraine medications (including ibuprofen or other NSAIDS) prior to study evaluation.
* Allergy to any of the medications used in our migraine regimen protocol.
* Patients exhibiting focal clinical neurological exam findings that the investigator deems makes the patient not a good candidate for this study.
* Patients with underlying abnormal brain pathology (e.g. mass or bleed) as the potential cause of the migraine

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Change in baseline pain score by a numerical self-reported visual analog pain score (VAS) | Baseline and 15 minutes after completion of intervention
  Pre-and post-intervention pain scores (0 to 10) by a numerical self-reported visual analog pain score (VAS)

SECONDARY OUTCOMES:
Duration of pain relief using the VAS pain scale | 2 to 6 days
  Data to be collected on this phone follow-up include return of migraine/headache using the VAS pain scale; return to ED or PMD for migraine/headache symptoms; and medications taken for headache since discharge from the ED.

CONTACTS AND LOCATIONS:
Overall Officials: Janice Sullivan, MD, Study Director — University of Louisville
Locations (2):
- United States (2):
  - Norton Children's Hospital, Louisville, Kentucky
  - Norton Children's Medical Center, Louisville, Kentucky

IPD SHARING:
Plan to Share IPD: No